CLINICAL TRIAL: NCT06092372
Title: The Role of Genetics in Weight Loss: a Randomized Diet Intervention Study in Individuals With High or Low Genetic Risk for Obesity (GENEROOS Study)
Brief Title: The Role of Genetics in Weight Loss
Acronym: GENEROOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Helsinki (Other)
Responsible Party: Principal Investigator, Andrea Ganna, Associate Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 945733HUS5832022
Record Dates: First submitted 2023-10-11; First posted 2023-10-23 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Body Mass Index (BMI)

STUDY DESIGN:
Masking Description: Participants were masked to their polygenic score group but not the diet intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Participants in the control group will be asked to fill out online surveys and book appointments for blood sample collection and weight measurements at the beginning and at the end of the study. In addition, participants will be asked to report their weight two more times during the study (in months 2 and 4) with an online survey that will be sent via the MyBiobank portal. The participation in the study ends with another personal visit to the clinic for blood sampling and weight measurement six months after registration. No other personal advice or support is provided to this group.
- Diet Intervention (Experimental): Participants in the diet intervention group will be asked to fill out online surveys and book appointments for blood sample collection and weight measurements at the beginning and at the end of the study. After visiting the clinic for the first time, each participant will be contacted to start a diet coaching program and to obtain an activity tracking device. In addition, each participant will be asked to report their weight two more times during the study (in months 2 and 4) with an online survey that will be sent to them via the online portal of the study (OmaBiopankki portal). The study participation ends with another personal visit to the clinic for blood sampling and weight measurement six months after registration.
  Interventions: Behavioral: Diet intervention program

INTERVENTIONS:
Behavioral: Diet intervention program — Participants will get 5 meals/day based on their calorie needs minus 500 kcal/day less than their daily calorie expenditure. All meals will be tracked via a mobile application, including any meals outside the recommended food plan. The calories will be calculated based on the information provided.
  To calculate the calories burned from any activities, all participants in the diet intervention arm will get an activity tracking device. The first calorie level is calculated based on the information in the registration form: age, height, weight, gender, and personal view of the daily activity. After that, and once the activity tracker is synced to the program, the calorie level is calculated based on the 7-day average calories burned.
  The external diet intervention provider will be blinded to whether the study participants belong to the top or bottom 5% of the polygenic score for BMI.
  Arms: Diet Intervention

SUMMARY:
The prevalence of both overweight and obesity is increasing at an alarming rate worldwide. In fact, it is estimated that 2.16 billion adults (38%) will be overweight and 1.12 billion adults (20%) will be obese by 2030. Among other risk factors (e.g., environmental, behavioral, and medical), genetics holds an important role. Genome-wide association studies have discovered hundreds of loci associated with body mass index (BMI). Polygenic scores (PS) are generated from a combination of millions of genetic variants that are associated with BMI. Several diet intervention studies aimed at reducing body weight in overweight and obese individuals. However, the effect of genetic background on the effectiveness of diet interventions is largely unknown. To our knowledge, the Diet Intervention Examining The Factors Interacting with Treatment Success (DIETFITS) trial is the only prospective study that has been designed to evaluate the effect of genotypes in modifying the impact of a healthy low-fat diet vs a healthy low-carbohydrate diet on weight change, but this study did not consider PS.

The aim of our study is to determine whether BMI PS impacts the effectiveness of dietary intervention in reducing BMI among individuals with elevated BMI.

To achieve this, the investigators will leverage the unique opportunity provided by the Finnish biobanks research environment to re-contact 1200 individuals who have extreme genetic predisposition for high/low BMI as measured by a PS for BMI and evaluate how a randomized diet intervention effect varies between the two extreme groups. In brief, the investigators will invite overweight (25-35 BMI) individuals with very high (Top 5%; n=600) and very low (Bottom 5%; n=600) PS for BMI. Half of the participants in each group will be subsequently randomized to enroll in a dietary/lifestyle coaching intervention program or the placebo group and not receive any dietary advice or information. All participants will be asked to answer an online questionnaire and provide a fasting blood sample at baseline and at the end of the study.

This well-powered prospective study leverages the unique opportunity to re-contact individuals at the extremes of BMI PS from a large pool of individuals with already available genetic information. This study will determine whether BMI PS can be used to identify overweight and obese individuals who are more likely to succeed in a reduced-energy dietary intervention, which will assist our efforts in curbing the overweight and obesity epidemic.

ELIGIBILITY:
Inclusion Criteria:

* 30-65 years old
* body mass index (BMI) of 25-35
* participants with genetic data available
* participants with a valid recontacting informed consent to their biobank

Exclusion Criteria:

* diagnosis of type I and II Diabetes Mellitus
* history of bariatric surgery
* diagnosis of schizophrenia and intellectual disability
* diagnosis of dementia and Parkinson's
* diagnosis of visual impairment
* diagnosis of multiple sclerosis
* pregnancy or breastfeeding during enrollment screening

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2024-11-08 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Interaction between the top and bottom 5th percentile of the polygenic score (PS) distribution for body mass index (BMI) distribution and BMI reduction | Six months
  The investigators will test the interaction between the BMI PS groups (i.e., top and bottom 5% PS for the BMI groups) and intervention groups (i.e. diet intervention and control) in their association with BMI differences between baseline and after 6 months (ΔBMI). More specifically, the investigators will test this interaction using a linear model such as ΔBMI ~ intervention_group*BMI_PS_group + age + age^2 + sex. In other words, the investigators will assess whether the effect of diet intervention on BMI reduction differs by the polygenic score for BMI among participants.
  BMI will be calculated based on the lab-measured body weight and height of each participant and according to the BMI calculation formula (i.e., weight in kilograms divided by height in meters squared).

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Ganna, Principal Investigator — University of Helsinki
Locations (1):
- Finnish Clinical Biobank Tampere, Tampere, Pirkanmaa, Finland

IPD SHARING:
Plan to Share IPD: No
Access to individual participant data can be obtained via FinnGenious (https://site.fingenious.fi/en/) and via study PI